CLINICAL TRIAL: NCT01759316
Title: Nasal Intermittent Positive Pressure Ventilation and Mechanical Ventilation With Heliox in Preterm Infants With Respiratory Distress Syndrome
Brief Title: Heliox in Preterm Infants With Respiratory Distress Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Yuan Shi, Director, Head of Pediatrics, Principal Investigator, Clinical Professor, Third Military Medical University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: Lixue
Record Dates: First submitted 2012-12-07; First posted 2013-01-03 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2013-10

CONDITIONS: Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — heliox

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- heliox (Active Comparator): Heliox is use in this group
  Interventions: Other: heliox
- Placebo (Placebo Comparator): Oxygen is used in this group
  Interventions: Other: heliox

INTERVENTIONS:
Other: heliox — heliox or oxygen is used in the two groups respectively

SUMMARY:
Heliox can lower respiratory resistance, improve the oxygenation, reduce respiratory distress and lung injury caused by mechanical ventilation.

DETAILED DESCRIPTION:
Heliox can improve the oxygenation, reduce respiratory distress and lung injury caused by mechanical ventilation.

Heliox has not been widely used. More studies on the effects and safety of Heliox in addition to NIPPV and mechanical ventilation should be tried.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age more than 28 weeks and less than 32 weeks
* Diagnosed as respiratory distress syndrome
* Need to use NIPPV ventilation
* No congenital diseases or hereditary diseases
* With an informed consent form

Exclusion Criteria:

* With congenital diseases or hereditary diseases
* Intubated in the delivery room
* Need surgery

Ages: 28 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2012-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
length of ventilation and risk of mechanical ventilation | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  The primary outcome is the length of ventilation and risk of mechanical ventilation of participants.

SECONDARY OUTCOMES:
Transcutaneous blood gas analysis，ventilator parameters and lung inflammation cytokines | participants will be followed for the duration of hospital stay, an expected average of 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Shi, MD, PhD, Study Chair — Dpartment of Pediatrics, Daping Hospital, Third Military Medical University
Locations (2):
- China (2):
  - Daping Hospital, China, Chongqing Municipality
  - Daping Hospital and Research Institute of Surgery, Chongqing